CLINICAL TRIAL: NCT02515643
Title: Estimating the Contribution of Renal Function to Endothelial Dysfunction by a Two-cohort Study: Living Kidney Donors and Their Transplant Recipients
Brief Title: Contribution of Renal Function to Endothelial Dysfunction in Living Kidney Donors and Transplant Recipients
Acronym: CONFUCIUS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Collaborators: Teva Pharmaceutical Industries, Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: PR(AG)219/2014
Record Dates: First submitted 2015-07-10; First posted 2015-08-05 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Disorder Related to Renal Transplantation; Chronic Kidney Disease; Endothelial Dysfunction
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Endothelial dysfunction in Cohort 1: Assessment of endothelial dysfunction in healthy subjects who will undergo a nephrectomy as part of the living donor program at each participating center.
  Interventions: Other: Endothelial dysfunction
- Endothelial dysfunction in Cohort 2: Assessment of endothelial dysfunction in renal transplant recipients from cohort 1
  Interventions: Other: Endothelial dysfunction

INTERVENTIONS:
Other: Endothelial dysfunction — One month before surgery and one year after, the following procedures will be performed in donors and recipients:
  1. Blood samples will be obtained for the measurement of endothelial dysfunction and low grade inflammation markers.
  2. Atherosclerotic burden: carotid ultrasound to determine the number of plaques and intima-media thickness, carotid-femoral pulse wave velocity (m/s) will be performed by pulse tonometry.
  3. Ambulatory blood pressure monitoring with overnight-automated ABPM monitor
  4. Estimation of glomerular filtration rate by Iohexol method

SUMMARY:
Endothelial dysfunction one-year after transplantation mainly depends on transplant-associated factors and only marginally on reduced renal function.

OBJETIVES Primary objective Estimate the contribution of renal dysfunction to endothelial dysfunction in two cohorts of patients, living kidney donors and their transplant recipients.

Secondary objectives

To evaluate in both cohorts of patients before and after nephrectomy/transplantation the evolution of the following parameters:

1. Renal function (iohexolGFR, proteinuria/microalbuminuria).
2. Blood pressure (24 h ambulatory blood pressure measurement)
3. Surrogate variables of subclinical atherosclerosis (carotid ultrasound, ankle-brachial index, pulse wave velocity).

DESIGN Non-interventional, prospective, multicenter, longitudinal study of two cohorts: living kidney donors and their transplant recipients.

DETAILED DESCRIPTION:
HYPOTHESIS

BACKGROUND: Chronic kidney disease (CKD) is associated with endothelial dysfunction, but the link between cardiovascular risk and CKD is difficult to establish because other conditions such as diabetes, hypertension and transplant-related factors are present in these patients. Living donors are healthy individuals that represent a near-ideal experimental model of CKD since they undergo a time-defined reduction of GFR after nephrectomy in the absence of other confounding factors present in patients with mild to moderate CKD.

HYPOTHESIS: Reduction of GFR after donation is associated with increased while renal transplantation is associated with reduced endothelial dysfunction markers.

AIM: To prospectively evaluate biomarkers of endothelial dysfunction and surrogate variables of subclinical atherosclerosis in a cohort of living kidney donors before and one year after donation and in their recipients before and one year after transplantation.

PATIENTS AND METHODS: In two cohorts of 60 living kidney donors (1 month before and 1 year after donation) and in their 60 renal transplant recipients (1 month before and 1 year after transplantation) the following variables will be recorded: iohexol glomerular filtration rate (GFR), proteinuria, microalbuminuria, insulinemia, oral glucose tolerance test, total and LDL/HDL cholesterol, number of carotid plaques and intima-media thickness, carotid-femoral pulse wave velocity, ankle-brachial index, 24-hours ambulatory monitoring of blood pressure. The following biomarkers of endothelial dysfunction and subclinical inflammation will be determined: SVCAM-1, PTX3, ICAM-1, von Willebrand factor, E-selectin, platelet/endothelial cell adhesion molecule (PECAM1), interleukin 6 (IL-6), soluble receptor of tumor necrosis factor (sTNFR1 and sTNFR2), high sensitive C reactive protein (hs-CRP) and soluble TNF-like weak inducer of apoptosis (sTWEAK).

EXPECTED RESULTS. In healthy subjects decrease of renal function after living donation will be associated with increased endothelial dysfunction markers. On the contrary, after transplantation a decrease of endothelial dysfunction markers will be observed. Despite at one year both cohorts of patients will have a similar GFR, the investigators expect that amelioration of endothelial dysfunction in transplants will be higher than worsening of endothelial dysfunction in their donors. Thus, the study of these two cohorts will allow estimating the contribution of renal dysfunction per se and transplant-associated comorbidities to endothelial dysfunction in chronic kidney disease.

ELIGIBILITY:
Inclusion Criteria cohort 1:

* No history of familiar nephropathies and/other diseases that may increase the risk for renal disease in the future.
* Donor age ≥ 18 years
* Isotopic GFR > 80 ml/min/1.73m2
* Microalbuminuria< 30 mg/g
* Normal urinary sediment
* Normal blood pressure defined as <120/90 mmHg and without other risk factors for cardiovascular disease, and with good/normal kidney function or well-controlled hypertension with one anti-hypertensive drug,
* No previous history of diabetes including gestational diabetes and fasting glucose < 126 mg/dl and 2h serum glucose after 75 g oral glucose tolerance test < 200 mg/dl
* Signed informed consent

Inclusion criteria cohort 2:

* Chronic kidney disease stage 5
* Negative complement dependent lymphocytotoxicity donor-recipient cross-match.
* Informed signed consent

Exclusion Criteria cohort 1:

* History of cancer except non-melanoma cutaneous neoplasia
* History of vasculitis (e.g. lupus), sarcoidosis, gastrointestinal inflammatory diseases, autoimmune-disease
* History of major cardiovascular events
* History of deep vein thrombosis or pulmonary embolism.
* Active infection including hepatitis B, C and HIV infections.
* Anatomic vascular variants precluding laparoscopic nephrectomy
* Renal stones except a solitary lithiasis< 1.5 cm once metabolic disorders are ruled out
* Major psychiatric disorders
* Active alcohol, tobacco or drug abuse
* Obesity defined as body mass index > 35 kg/m2.
* Pregnancy

Exclusion criteria cohort 2:

* Glomerulonephritis with high recurrence rate after transplantation (focal segmental glomerulosclerosis and type II membranoproliferative glomerulonephritis)
* Severe aortoiliac atherosclerosis precluding transplantation
* Major psychiatric disorders
* Alcohol and drug abuse
* Active infection
* Patients requiring desensitization treatment before transplantation.
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cohort 1
  Healthy subjects who will undergo a nephrectomy as part of the living donor program at each participating center.
  Cohort 2
  Renal transplant recipients from cohort 1
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2015-07; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Percentual change of sVCAM | 1 year
  Biomarker of endothelial dysfunction: Soluble VCAM (vascular cell adhesion molecule). Determination of serum levels by Luminex. Percentual change between baseline and 1 year levels.

SECONDARY OUTCOMES:
Glomerular filtration rate | 1 year
  Renal function will be estimated before donation by iohexol clearance and expressed as mL/min/1.73 m2 in donors and at 1 year in donors and recipients.
Microalbuminuria | 1 year
  Microalbuminuria (mg/g creatinine) will be determined before donation and at 1 year in donors and at 1 year in transplant recipients.
Blood pressure (24 h ambulatory blood pressure measurement) | 1 year
  Ambulatory blood pressure monitoring (mm Hg) with overnight-automated ABPM monitor (Spacelab 90207; Spacelabs Healthcare,USA) with appropriate cuff sizes for each patient.
Number of carotid plaques and carotid intima-media thickness | 1 year
  Atherosclerotic burden: carotid ultrasound to determine the number of plaques and intima-media thickness will be held in both carotid arteries with a high-frequency (8-12 MHz) linear transducer (ESAOTE, 7300, Florence, Italy),
Pulse wave velocity. | 1 year
  Carotid-femoral pulse wave velocity (m/s) will be measured by pulse tonometry (Sphingmocor Atcor, EM3, Australia).
Percentual change of sICAM | 1 year
  Biomarker of endothelial dysfunction: Soluble ICAM (intercellular adhesion molecule). Determination of serum levels by Luminex. Percentual change between baseline baseline and 1 year levels.
Percentual change of PECAM | 1 year
  Biomarker of endothelial dysfunction: PECAM (platelet/endothelial cell adhesion molecule). Determination of serum levels by Luminex. Percentual change between baseline baseline and 1 year levels.
Percentual change of vWF | 1 year
  Biomarker of endothelial dysfunction: vWF (von Willebrand factor). Determination of serum levels by Luminex. Percentual change between baseline baseline and 1 year levels.
Percentual change of E-selectin | 1 year
  Biomarker of endothelial dysfunction: Soluble E-selectin. Determination of serum levels by Luminex.Percentual change between baseline baseline and 1 year levels.
Percentual change of PTX3 | 1 year
  Biomarker of endothelial dysfunction: PTX3 (pentraxin). Determination of serum levels by ELISA. Percentual change between baseline baseline and 1 year levels.
Percentual change of hs-CRP | 1 year
  Biomarker of subclinical inflammation: hs-CRP (high sensitive C reactive protein). Determination of serum levels by nephelometry. Percentual change between baseline baseline and 1 year levels.
Percentual change of IL-6 | 1 year
  Biomarker of subclinical inflammation: IL-6 IL-6 (interleukin 6). Determination of serum levels by Luminex. Percentual change between baseline baseline and 1 year levels.
Percentual change of sTNFR1 and sTNFR2 | 1 year
  Biomarker of subclinical inflammation: sTNFR1 and sTNFR2 (soluble tumor necrosis factor receptor). Determination of serum levels by Luminex. Percentual change between baseline baseline and 1 year levels.
Percentual change of sTWEAK | 1 year
  Biomarker of subclinical inflammation: sTWEAK (soluble TNF-like weak inducer of apoptosis). Determination of serum levels by ELISA. Percentual change between baseline baseline and 1 year levels.

CONTACTS AND LOCATIONS:
Overall Officials: Francesc Moreso, MD, PhD, Principal Investigator — Hospital Vall d'Hebron
Locations (4):
- Spain (4):
  - Hospital del Mar, Barcelona, Barcelona
  - Vall d'Hebron Research Institute, Barcelona, Barcelona
  - Hospital Universitario Canarias, Santa Cruz de Tenerife, Canary Islands
  - Hospital Regional Universitario Carlos Haya, Málaga, Malaga